CLINICAL TRIAL: NCT03399227
Title: Skeletal Effects of Liver Transplantation
Brief Title: Liver Transplantation: Skeletal Effects
Status: Withdrawn | Type: Observational
Why Stopped: no funding
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Katharina Kerschan-Schindl, MD, Assoc professor, Medical University of Vienna
Other Study IDs: 1713/2017
Record Dates: First submitted 2018-01-05; First posted 2018-01-16 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Liver Diseases; Transplant-Related Disorder; Osteoporosis
Keywords: Bone microarchitecture
MeSH Terms: conditions — Liver Diseases; Osteoporosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — venous blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Liver transplantation recipients: Venipuncture (6x) Bone mineral density measurement: lumbar spine, hip region (3x) high resolution peripheral quantitative CT: radius, tibia (3x)
- Control group: Venipuncture (1x) Bone mineral density measurement: lumbar spine, hip region (1x) high resolution peripheral quantitative CT: radius, tibia (1x)

SUMMARY:
Fifty patients awaiting liver transplantation and 50 age and gender matched control subjects with normal liver function will be included in the study. The aim of this project is to compare liver transplantation recipients'bone microarchitecture with healthy controls and to evaluate patients' changes within one year after transplantation

DETAILED DESCRIPTION:
Background: Solid organ transplantation recipients have a high prevalence of osteoporosis and fragility fractures. Deteriorated bone architecture has been shown by high resolution computed tomography (HR-pQCT) in kidney and lung transplantation recipients. In liver transplantation (LeTx) recipients, bone microarchitecture has only been evaluated using the trabecular bone score in a retrospective cohort study; a degraded or partially degraded microarchitecture was detected in most of the patients.

Aim: The aim of this project is to compare LeTx recipients' bone microarchitecture with healthy controls and to evaluate patients' changes within one year after transplantation.

Methods: HR-pQCT scans of the distal radius and tibia as well as areal bone mineral density measurement of the lumbar spine and hip region will be performed before Tx, 1 and 12 months after Tx in 50 patients. Anabolic and catabolic markers of bone turnover (sclerostin, dickkopf 1, periostin) and traditional bone turnover markers will be evaluated preoperatively, on the day of surgery, and 4 times within the first year after LeTx. In healthy age- and sex-matched controls HR-pQCT, bone mineral density and laboratory parameters will be assessed once.

Hypotheses: Based on the HR-pQCT data of kidney and lung transplantation recipients and the trabecular bone score of LeTx recipients, the investigators hypothesize that LeTX recipients have deteriorated bone microarchitecture.

Expected outcome: Since bone fragility is not only determined by BMD but bone architecture as well, HR-pQCT data give important information on the patients' bone fragility. The knowledge of the course of bone microarchitecture after liver transplantation may help to develop strategies preventing fragility fractures in LeTx recipients.

ELIGIBILITY:
Inclusion Criteria:

* Women, men awaiting liver Transplantation
* 20-70 years of age

Exclusion Criteria:

* Subjects with a history of prior solid organ transplantation
* Subjects awaiting a combined liver-kidney transplantation
* Cancer within the previous 5 years - except for hepatocellular carcinoma, neuroendocrine tumors and hemangioendothelioma with indication for liver transplantation
* Rheumatoid arthritis
* Severe renal insufficiency (chronic kidney disease IV, V)
* Immobilisation
* Intake of drugs with potential effects on BMD like lithium, estrogen-replacement therapy, selective Estrogen-receptor modulators, oral bisphosphonates in the last three months, denosumab and parenteral bisphosphonates in the last year - except calcium, vitamin D and medication necessary for the underlying disease
* Non-osteoporotic bone disease
* Recent fragility fracture within 6 months

Control group:

Inclusion Criteria:

* Women, men
* 20-70 years of age
* Normal liver function (defined as liver function parameters and transaminases, such as albumin, thromboplastin time, alanine-aminotransferase, aspartate-aminotransferase, and gamma-glutamyl-transferase within the normal range)

Additional exclusion Criteria:

* Osteoporosis according to BMD measurement or osteopenia plus fragility fracture
* Liver disease (defined as evidence of significant liver disease according to laboratory testing)

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 50 patients awaiting liver transplantation and 50 age and gender matched healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Bone microarchitecture of the distal radius | 12 months to posttransplantation
  trabecular bone mineral density measurement (XCT)

SECONDARY OUTCOMES:
Bone microarchitecture of the distal radius | pretransplantation to 12 after transplantation
  bone volume fraction (%)
Bone microarchitecture of the distal radius | pretransplantation to 12 after transplantation
  trabecular homogeneity (mm)
Bone microarchitecture of the distal radius | pretransplantation to 12 after transplantation
  trabecular number (mm-1)
Bone microarchitecture of the distal radius | pretransplantation to 12 after transplantation
  trabecular thickness (mm)
Bone microarchitecture of the distal radius | pretransplantation to 12 months after transplantation
  trabecular separation (mm)

OTHER OUTCOMES:
Bone mineral density | pretransplantation to 12 after transplantation
  areal bone density measurement of the lumbar spine (T score)
Bone mineral density | pretransplantation to 12 after transplantation
  areal bone density measurement of the hip region (T score)
Biochemical | pretransplantation to 12 after transplantation
  Serum levels of osteocalcin
Biochemical | pretransplantation to 12 after transplantation
  Serum levels of bone-specific alkaline phosphatase
Biochemical | pretransplantation to 12 after transplantation
  Serum levels of procollagen type 1 amino-terminal propeptide
Biochemical | pretransplantation to 12 after transplantation
  Serum levels of tartrate resistant acid phosphatase
Biochemical | pretransplantation to 12 after transplantation
  Serum levels of carboxy-terminal collagen crosslinks
Biochemical | pretransplantation to 12 after transplantation
  Serum levels of dickkopf 1
Biochemical | pretransplantation to 12 after transplantation
  Serum levels of periostin
Biochemical | pretransplantation to 12 after transplantation
  Serum levels of sclerostin

CONTACTS AND LOCATIONS:
Overall Officials: Katharina Kerschan-Schindl, MD, Principal Investigator — Medical University of Vienna

IPD SHARING:
Plan to Share IPD: Undecided